CLINICAL TRIAL: NCT02859506
Title: Eating Behaviour and Gustatory Sensitivity Before and After Liver Transplant in Cirrhotic Patients
Acronym: GREFFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BRONDEL INRA 2013
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Eating Behaviour; Liver Transplant
MeSH Terms: conditions — Feeding Behavior

ARMS (4):
- liver transplant (Experimental)
  Interventions: Other: Respiratory quotient; Other: Olfactory liking
- kidney transplant (Active Comparator)
  Interventions: Other: Respiratory quotient; Other: Olfactory liking
- control (Placebo Comparator)
  Interventions: Other: Respiratory quotient; Other: Olfactory liking
- stable liver damage (Active Comparator)
  Interventions: Other: Respiratory quotient; Other: Olfactory liking

INTERVENTIONS:
Other: Respiratory quotient
Other: Olfactory liking

SUMMARY:
Today, we know that olfactogustatory alterations occur in cirrhotic patients before the liver transplant but no study has been conducted to show eventual disturbances after the transplantation able to explain modifications in eating behaviour. In parallel, the metabolic status, itself dependent on liver metabolism, influences food preferences and is modified after the transplantation as the liver recovers its ability to store glycogen, but is not able to inform the brain as the afferent nerve impulses have been suppressed. The innovative aspect of this project is to provide information on the importance of the liver in the regulation of energy homeostasis.

The results of this study will improve our understanding of eating behaviour and olfactogustatory sensitivity and allow us to orient liver transplant patients towards appropriate diets.

ELIGIBILITY:
Inclusion Criteria:

* persons who have provided written informed consent
* persons aged between 18 and 70 years
* persons waiting for a liver transplantation (group LT)
* persons with stable liver damage
* persons waiting for a kidney transplantation (KT)
* healthy subjects (control group) no known disease

Exclusion Criteria:

* persons without national health insurance cover
* persons with chronic infection,
* persons with acute infection,
* persons with progressive cancer,
* persons with an antibiotic treatment,
* persons who drink alcohol,
* pregnant or breast-feeding women,
* persons with an aversion to the foods proposed in the study,
* persons taking treatments known to interfere with gustatory and olfactory performance,
* adults under guardianship

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-07-03 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Change in respiratory quotient (RQ) by indirect calorimetry compared with baseline values | At month 0, month 3, month 9 and month 15
Change in olfactory liking compared with baseline values by questionnaire | At month 0, month 3, month 9 and month 15

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Dijon, France